CLINICAL TRIAL: NCT06799143
Title: Follow-up Evaluation of Osteoporotic Women Who Underwent a Local Osteo-Enhancement Procedure (LOEP) in the Proximal Femur
Brief Title: Copley II: Long-term Outcome Follow-up Study of Osteoporotic Women Who Underwent a Local Osteo-Enhancement Procedure (LOEP) in the Proximal Femur
Status: Completed | Type: Observational
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PRE-US-101.0
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Osteopenic Women; Proximal Femur Fracture
Keywords: LOEP; osteoporosis; femur fracture
MeSH Terms: conditions — Proximal Femoral Fractures; Osteoporosis; Femoral Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate longer-term (5-7 years) outcomes of the twelve (12) subjects treated with AGN1 Femoral LOEP in the clinical study "A Prospective Pilot Evaluation of Percutaneous Osteo-supplementation in the Proximal Femur of Osteoporotic Patients". Performance will be evaluated via medical history evaluation, X-ray, DXA, CT and mobility testing.

The study will look at the extent to which the benefits demonstrated in the initial, baseline study were sustained over time. In this manner, it may be possible to determine the rate of change in BMD following the treatment; thereby allowing prediction of the total benefit period. In addition, this longer period of observation allows for further evaluation of the safety profile of the material in osteoporosis patients.

DETAILED DESCRIPTION:
This observational single arm study will be broken into two parts:

1. A retrospective component which will evaluate the original FRAX score along with any events or medications received after the end of the original study.
2. A prospective component which will evaluate longer term outcomes following the use of the AGN1 synthetic bone graft material in a local osteoenhancement procedure through evaluation of mobility and imaging.

In the original study, subjects completed a twenty-four (24) month follow-up visit after receiving a unilateral hip injection with the device. The contralateral hip acted as the control. The purpose of the study was to determine the safety of the injection as well as the initial improvement in femoral bone density in a twenty-four (24) month period.

In this follow-up study the subjects, after signing the informed consent form, will complete a short medical history (focused on their osteoporosis management) and a mobility test.

Subjects will also undergo a DXA, X-ray and CT scans of both hips.

ELIGIBILITY:
Inclusion Criteria:

* participated in the original study and signed the consent form
* received treatment with AGN1 Femoral LOEP
* completed the study.

Exclusion Criteria:

* There is no exclusion criteria for this study.

Min Age: 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Females aged 56 or older and menses have ceased for at least one year. Subjects that were participants in the original study that signed a consent form, received treatment with AGN1 Femoral LOEP and completed the original study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | through study completion, an average of 30 days
  Bone mineral density (BMD) assessed by DXA scans (T-score ) of the treated hip compared to nontreated hip (femoral neck).
Bone Mineral Density | through study completion, an average of 30 days
  Bone mineral density (BMD) assessed by DXA scans (absolute value measurement) of the treated hip compared to nontreated hip (femoral neck).
Bone Mineral Density | through study completion, an average of 30 days
  Percent change compared to baseline for the treated femoral neck measurement of BMD.
Bone Mineral Density | through study completion, an average of 30 days
  Percent change compared to baseline for the untreated femoral neck measurement of BMD.
Bone Mineral Density | through study completion, an average of 30 days
  Bilateral hip CT scan analysis of the trabecular bone density.
Bone Mineral Density | through study completion, an average of 30 days
  Bilateral hip CT scan analysis of the trabecular bone volume.
Bone Mineral Density | through study completion, an average of 30 days
  Bilateral hip CT scan analysis of the cortical bone density.
Bone Mineral Density | through study completion, an average of 30 days
  Bilateral hip CT scan analysis of the cortical bone volume.
Bone Mineral Density | through study completion, an average of 30 days
  Bilateral hip CT scan analysis of any qualitative observations compared to baseline CT scans.

SECONDARY OUTCOMES:
Subject Interview | through study completion, an average of 30 days
  All osteoporosis related events (as defined by the Investigator) from the twenty-four (24) month follow-up visit to current point-in-time including fragility fractures, changes in mobility and medication reactions.
Subject Interview | through study completion, an average of 30 days
  All osteoporosis medication use including vitamins and supplements from the twenty-four (24) month follow-up visit to current point-in-time.
Subject Interview | through study completion, an average of 30 days
  Any physical activity/exercise program from the twenty-four (24) month follow-up visit to current point-in-time.
FRAX Index Risk Assessment | through study completion, an average of 30 days
  Comparative calculation of a FRAX index for hip fracture risk based on BMD data from the treatment and contralateral hip using pre-procedure data compared to current point-in-time.